CLINICAL TRIAL: NCT03061708
Title: Phase II Trial of Single Agent AZD2014 in RICTOR Amplified or Over-expressed GC Patients as Second-line Therapy
Brief Title: Trial of Single Agent AZD2014 in RICTOR Amplified GC Patients as Second-line Therapy
Acronym: AZD2014
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of efficacy
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeeyun Lee, professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-08-001
Record Dates: First submitted 2017-02-10; First posted 2017-02-23 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms | interventions — vistusertib

STUDY DESIGN:
Intervention Model Description: AZD2014 50mg BD continuous schedule of a 28 day cycle
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AZD2014 50mg BD continuous schedule of a 28 day cycle (Experimental): AZD2014 50mg BD continuous schedule of a 28 day cycle
  Interventions: Drug: AZD2014

INTERVENTIONS:
Drug: AZD2014 — mTOR inhibitor

SUMMARY:
Phase II trial of AZD2014 in RICTOR amplified or overexpressed GC patients as second-line chemotherapy AZD2014 50mg BD continuous schedule of a 28 day cycle

DETAILED DESCRIPTION:
Tumour evaluation using RECIST 1.1 will be conducted at screening (within 28 days prior to first dose) and every 8 weeks relative to the date of first dose, up to week 40, then every 16 weeks until objective disease progression (within a window of +/- 7 days of the scheduled date).

Study treatment will be continued until objective disease progression (unless other criteria for 3 treatment discontinuation are met). Patients may continue AZD2014 beyond progression (according to RECIST 1.1), at the discretion of the investigator if they are clinically benefiting from the treatment and they do not meet any other discontinuation criteria.

If a patient discontinues study treatment prior to disease progression, they should continue to be assessed using RECIST 1.1 until disease progression and then followed up for survival.

Assessments for survival should be made every 8 weeks following objective disease progression. The details of first and subsequent therapies for cancer, after discontinuation of treatment, will be collected. The imaging modalities used for RECIST 1.1 assessment will be CT or MRI scans of chest, abdomen and pelvis. RECIST 1.1 scans will be analysed by the investigator on site.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of fully informed consent prior to any study specific procedures.
2. Patients must be ≥20 years of age.
3. Advanced gastric adenocarcinoma (including GEJ) that has progressed during or after firstline therapy.
4. Previous adjuvant/neoadjuvant chemotherapy is allowed, if completed more than 6 months prior to starting the 1st line therapy.
5. Provision of tumor sample (from either a resection or biopsy)
6. Patients with RICTOR amplification or overexpression through the VIKTORY trial.
7. Patients are willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.
8. ECOG performance status 0-2.
9. Patients must have a life expectancy ≥ 3 months from proposed first dose date.
10. Patients must have acceptable bone marrow, liver and renal function -
11. At least one measurable lesion that can be accurately assessed by imaging or physical examination at baseline and following up visits.
12. Negative urine or serum pregnancy test within 28 days of study treatment, confirmed prior to treatment on day 1.

Exclusion Criteria:

1. More than one prior chemotherapy regimen for the treatment of gastric cancer in the advanced setting.
2. Any previous treatment with PIK3CA, AKT or mTOR inhibitor or agents with mixed PI3K / mTOR activity.
3. Patients with second primary cancer,
4. Patients unable to swallow orally administered medication.
5. Previous major surgery within 4weeks prior to enrollment.
6. For AZD2014: Exposure to potent or moderate inhibitors or inducers of CYP3A4/5 if taken within the stated washout periods before the first dose of study treatment Inhibitors
7. Exposure to potent or moderate inhibitors or inducers of CYP2C8 if taken within the stated washout periods before the first dose of study treatment
8. With the exception of alopecia, any ongoing toxicities (>CTCAE grade 1) caused by previous cancer therapy.
9. Intestinal obstruction or CTCAE grade 3 or grade 4 upper GI bleeding within 4 weeks before the enrollment.
10. Resting ECG with measurable QTcB > 450 msec on 2 or more time points within a 24 hour period or family history of long QT syndrome.
11. Patients with cardiac problem
12. Active or untreated brain metastases or spinal cord compression Patients with treated brain metastases or spinal cord compression are eligible if they have minimal neurologic symptoms, evidence of stable disease (for at least 1 month) or response on follow-up scan, and require no corticosteroid therapy for ≥ 1 week.
13. Female patients who are breast-feeding or child-bearing
14. Any evidence of severe or uncontrolled systemic disease, active infection, active bleeding diatheses or renal transplant, including any patient known to have hepatitis B, hepatitis C or human immunodeficiency virus (HIV)
15. Patients with proteinuria (3+ on dipstick analysis )

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-11-16 (Actual); Study Completion 2018-11-16 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) by RECIST 1.1 | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeeyun Lee, Md,PhD, Principal Investigator — SamsungMedicalCenter
Locations (1):
- Samsung Medical Center, Seoul, South Korea